CLINICAL TRIAL: NCT01149057
Title: An Open-Label Study to Evaluate the Efficacy and Safety Of Tocilizumab in Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to Current Non-biologic DMARDs and/or Biologic DMARDs
Brief Title: A Study of RoActemra/Actemra (Tocilizumab) in Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to Current Non-Biologic and/or Biologic DMARDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Clalit Health Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22873
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg intravenously, every 4 weeks for 96 weeks

SUMMARY:
This single arm, open-label study will evaluate the efficacy and safety of RoActemra/Actemra (tocilizumab) in patients with active, moderate to severe rheumatoid arthritis who have an inadequate response to non-biologic and/or biologic disease-modifying antirheumatic drugs (DMARDs). Patients will receive intravenous RoActemra/Actemra at a dose of 8 mg/kg every 4 weeks. Anticipated time on study treatment is 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Active moderate to severe rheumatoid arthritis
* Inadequate response to >/=3 DMARDs (non-biologic and/or biologic)
* Current treatment at stable dose for >/=8 weeks
* Etanercept discontinued >/=2 weeks, Anakinra >/=1 week, Infliximab, Adalimumab, Abatacept, Golimumab, Certolizumab >/=4 weeks, prior to baseline visit. Patients have discontinued MabThera/Rituxan or Ocrelizumab >/=16 weeks, and must have proven B-cell repletion

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following baseline
* Rheumatic autoimmune disease other than RA
* Functional class IV (American College of Rheumatology Classification)
* Prior history or current inflammatory joint disease other than RA
* Oral corticosteroids at a dose of >10 mg/day prednisone equivalent
* Positive hepatitis B surface antigen (HBsAg) and / or total hepatitis B core antibodies (HBcAb) or hepatitis C virus (HCV) antibody
* Current or history of recurrent bacterial, viral, fungal or mycobaterial infection
* History of or currently active primary or secondary immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2010-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- Israel (13):
  - Afula
  - Ashkelon
  - Beer Yaakov
  - Beersheba
  - Hadera
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Tel Aviv

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Participants received tocilizumab 8 milligrams per kilograms (mg/kg) intravenous (IV) infusion every 4 weeks for a period of 96 weeks.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 145
Completed | 88
Not Completed | 57
Not completed — Lack of Efficacy | 16
Not completed — Adverse Event | 13
Not completed — Withdrawal by Subject | 9
Not completed — Positive Hepatitis B Core Antibody | 5
Not completed — B Cell Depletion | 4
Not completed — Participant Non-Compliance | 2
Not completed — Lost to Follow-up | 1
Not completed — High Parathyroid Hormone Value | 1
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population: all participants who have received any part of an infusion of the study drug.
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg IV infusion every 4 weeks for a period of 96 weeks.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (13.4)
Gender [Count of Participants; unit: Participants]
  Female | 121
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Score at Week 24 in Intent-to-treat (ITT) Population
Description: The FACIT-Fatigue score was calculated according to a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worst score) to 52 (best score).
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analysed=participants with available data for this endpoint. Here, 'n' signifies participants with available data at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 142
units on a scale
  Baseline (n=142) | 21.2 (11.8)
  Change From Baseline at Week 24 (n=118) | 5.4 (9.6)
Statistical Analysis 1: Comparison: Tocilizumab; Analysis was performed using paired sample t-test for change from baseline; Test type: Superiority or Other; p < 0.0001, Paired sample T-test

2. Secondary Outcome: Change From Baseline in Bone Mineral Density (BMD) in Lumbar Spine, Total Hip and Femoral Neck Regions at End of Study
Description: BMD was measured by dual energy X-ray absorptiometry (DXA) and T-scores (a standard deviation [SD] compared with the peak BMD value of an adult aged from 20 to 30 years) were calculated. Osteopenia was defined by a T-score between -1 and -2.5 SD and osteoporosis as a T-score below -2.5 SD, according to the World Health Organization (WHO) guidelines. T-scores for L1-L4 lumbar spine, total spine, total hip (left), and femoral neck (left) were calculated.
Time Frame: Baseline, End of the study (up to Week 100)
Population: ITT population. Number of participants analyzed=participants with available data for this endpoint. Here, 'n' signifies the number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Tocilizumab
Number analyzed (Participants) | 137
T-score
  L1-L4: Baseline (n=40) | -0.81 (1.35)
  L1-L4: Change From Baseline at End (n=22) | -0.05 (0.39)
  Total Spine: Baseline (n=109) | -1.13 (1.33)
  Total Spine: Change From Baseline at End (n=65) | 0.04 (0.50)
  Total Hip-Left: Baseline (n=124) | -0.67 (1.16)
  Total Hip-Left: Change From Baseline at End (n=76) | 0.10 (0.37)
  Neck-Left: Baseline (n=137) | -1.11 (1.17)
  Neck-Left: Change From Baseline at End (n=85) | -0.05 (0.36)
Statistical Analysis 1: Comparison: Tocilizumab; Comparison of L1-L4 T-scores; Test type: Superiority or Other; p = 0.3778, ANCOVA — P value by analysis of covariance (ANCOVA) for the change from baseline, adjusted to number of days between the first and the second DXA test
Statistical Analysis 2: Comparison: Tocilizumab; Comparison of Total spine T-score; Test type: Superiority or Other; p = 0.1541, ANCOVA — P value by ANCOVA for the change from baseline, adjusted to number of days between the first and the second DXA test
Statistical Analysis 3: Comparison: Tocilizumab; Comparison of Total hip - left T-score; Test type: Superiority or Other; p = 0.7890, ANCOVA — P value by ANCOVA for the change from baseline, adjusted to number of days between the first and the second DXA test
Statistical Analysis 4: Comparison: Tocilizumab; Comparison of Femoral neck - left T-scores; Test type: Superiority or Other; p = 0.7094, ANCOVA — P value by ANCOVA for the change from baseline, adjusted to number of days between the first and the second DXA test

3. Secondary Outcome: Number of Participants Achieving Remission According to Disease Activity Score 28 (DAS28) at Weeks 24, 48, 72, and 96
Description: Remission was defined as DAS28 score less than (<) 2.6. The DAS28 score was a measure of the participant's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity (visual analog scale [VAS]: 0=no disease activity to 100=maximum disease activity) and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. In case of missing ESR value, C-Reactive Protein (CRP) was used to calculate DAS28. Higher scores represented higher disease activity.
Time Frame: Weeks 24, 48, 72 and 96
Population: ITT population. Number of participants analyzed=participants with available data for this endpoint. Here, 'n' signifies the number participants with available data for specified category.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 115
participants
  Week 24 (n=115) | 35
  Week 48 (n=95) | 37
  Week 72 (n=73) | 27
  Week 96 (n=72) | 33

4. Secondary Outcome: Percentage of Participants Achieving Remission According to DAS28 at Weeks 24, 48, 72, and 96
Description: Remission was defined as DAS28 score <2.6. The DAS28 score was a measure of the participant's disease activity calculated using the TJC [28 joints], SJC [28 joints], patient's global assessment of disease activity (VAS: 0=no disease activity to 100=maximum disease activity) and the ESR for a total possible score of 0 to approximately 10. In case of missing ESR value, CRP was used to calculate DAS28. Higher scores represented higher disease activity.
Time Frame: Weeks 24, 48, 72 and 96
Population: ITT population. Number of participants analyzed=participants with available data for this endpoint. Here, 'n' signifies number of participants with available data for specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 115
percentage of participants
  Week 24 (n=115) | 30.4
  Week 48 (n=95) | 38.9
  Week 72 (n=73) | 37.0
  Week 96 (n=72) | 45.8

5. Secondary Outcome: Percentage of Participants With DAS28 Good or Moderate European League Against Rheumatism (EULAR) Response at Weeks 24, 48, 72 and 96
Description: The DAS28 score was a measure of the participant's disease activity calculated using the TJC [28 joints], SJC [28 joints], patient's global assessment of disease activity (VAS: 0=no disease activity to 100=maximum disease activity) and the ESR for a total possible score of 0 to approximately 10. In case of missing ESR value, CRP was used to calculate DAS28. Higher scores represented higher disease activity. EULAR Good response: DAS28 ≤3.2 and a change from Baseline <-1.2. EULAR Moderate response: DAS28 greater than (>) 3.2 to less than or equal to (≤) 5.1 or a change from Baseline <-0.6 to greater than or equal to (≥) -1.2.
Time Frame: Weeks 24, 48, 72 and 96
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 114
percentage of participants
  Week 24 (n=114) | 94.8
  Week 48 (n=94) | 94.7
  Week 72 (n=73) | 90.4
  Week 96 (n=72) | 94.5

6. Secondary Outcome: Percentage of Participants Achieving Remission and Low Disease Activity According to Simplified Disease Activity Index (SDAI) at Weeks 24, 48, 72, and 96
Description: SDAI was calculated by a simple numerical sum of tender and swollen joint count (based on a 28-joint assessment), patient and physician global assessment of disease activity (VAS 0-10 centimeter [cm]), and level of CRP. SDAI total score 0-86; higher scores = greater effect due to disease activity. Remission was defined as SDAI score ≤3.3. Low disease activity was defined as SDAI score ≤11.0.
Time Frame: Weeks 24, 48, 72 and 96
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 107
percentage of participants
  Remission at Week 24 (n=107) | 10.3
  Low Disease Activity at Week 24 (n=107) | 41.1
  Remission at Week 48 (n=86) | 11.6
  Low Disease Activity at Week 48 (n=86) | 39.5
  Remission at Week 72 (n=60) | 16.7
  Low Disease Activity at Week 72 (n=60) | 51.7
  Remission at Week 96 (n=72) | 13.9
  Low Disease Activity at Week 96 (n=72) | 44.5

7. Secondary Outcome: Percentage of Participants Achieving Remission and Low Disease Activity According to Clinical Disease Activity Index (CDAI) at Weeks 24, 48, 72, and 96
Description: CDAI was calculated by a simple numerical sum of tender and swollen joint count (based on 28-joint assessment) and the patient and physician global disease assessment (VAS 0-10 cm). CDAI total score 0-76; higher scores = greater effect due to disease activity. Remission was defined as CDAI score ≤2.8. Low disease activity was defined as CDAI score ≤10.0.
Time Frame: Weeks 24, 48, 72 and 96
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 120
percentage of participants
  Remission at Week 24 (n=120) | 6.7
  Low Disease Activity at Week 24 (n=120) | 37.5
  Remission at Week 48 (n=97) | 9.3
  Low Disease Activity at Week 48 (n=97) | 36.1
  Remission at Week 72 (n=75) | 10.7
  Low Disease Activity at Week 72 (n=75) | 42.7
  Remission at Week 96 (n=80) | 17.5
  Low Disease Activity at Week 96 (n=80) | 47.5

8. Secondary Outcome: Change From Baseline in TJC At Weeks 24, 48, 72, and 96
Description: 68 joints are assessed for tenderness and joints are classified as tender/not tender giving a total possible tender joint count score of 0 to 68. A negative change from baseline indicated improvement.
Time Frame: Baseline; Weeks 24, 48, 72 and 96
Population: ITT population. Here, 'n' signifies the number of participants with available data at specified timepoints.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 145
tender joints
  Baseline (n=145) | 22.8 (14.2)
  Change From Baseline at Week 24 (n=124) | -13.4 (13.5)
  Change From Baseline at Week 48 (n=99) | -15.2 (13.4)
  Change From Baseline at Week 72 (n=79) | -13.9 (14.5)
  Change From Baseline at Week 96 (n=84) | -14.5 (12.4)
Statistical Analysis 1: Comparison: Tocilizumab; Change from baseline at Week 24; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: Tocilizumab; Change from baseline at Week 48; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test
Statistical Analysis 3: Comparison: Tocilizumab; Change from baseline at Week 72; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test
Statistical Analysis 4: Comparison: Tocilizumab; Change from baseline at Week 96; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test

9. Primary Outcome: Change From Baseline in FACIT Fatigue Score at Week 48 in ITT Population
Description: as for outcome 1
Time Frame: Baseline, Week 48
Population: ITT population. Number of participants analyzed=participants with available data at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 97
units on a scale | 6.7 (10.5)
Statistical Analysis 1: Comparison: Tocilizumab; Test type: Superiority or Other; p < 0.0001, Paired sample T-test

10. Primary Outcome: Change From Baseline in FACIT Fatigue Score at Week 72 in ITT Population
Description: as for outcome 1
Time Frame: Baseline, Week 72
Population: ITT population. Number of participants analyzed=participants with available data at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 75
units on a scale | 7.1 (10.7)
Statistical Analysis 1: Comparison: Tocilizumab; Test type: Superiority or Other; p < 0.0001, Paired sample T-test

11. Primary Outcome: Change From Baseline in FACIT Fatigue Score at Week 96 in ITT Population
Description: as for outcome 1
Time Frame: Baseline, Week 96
Population: ITT population. Number of participants analyzed=participants with available data at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 83
units on a scale | 7.3 (10.4)
Statistical Analysis 1: Comparison: Tocilizumab; Test type: Superiority or Other; p < 0.0001, Paired sample T-test

12. Primary Outcome: Change From Baseline in FACIT Fatigue Score at Week 24 in Per Protocol (PP) Population
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: Per Protocol (PP) population: all participants who completed the study. Number of participants analyzed=participants with available data for this outcome. Here 'n' signifies the participants with available data for specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 86
units on a scale
  Baseline (n=86) | 20.9 (10.9)
  Change From Baseline at Week 24 (n=80) | 5.0 (9.7)
Statistical Analysis 1: Comparison: Tocilizumab; Analysis was performed using paired sample t-test for change from baseline; Test type: Superiority or Other; p < 0.0001, Paired sample T-test

13. Primary Outcome: Change From Baseline in FACIT Fatigue Score at Week 48 in PP Population
Description: as for outcome 1
Time Frame: Baseline, Week 48
Population: Per Protocol (PP) population. Number of participants analyzed=participants with available data for specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 81
units on a scale | 6.8 (10.5)
Statistical Analysis 1: Comparison: Tocilizumab; Test type: Superiority or Other; p < 0.0001, Paired sample T-test

14. Primary Outcome: Change From Baseline in FACIT Fatigue Score at Week 72 in PP Population
Description: as for outcome 1
Time Frame: Baseline, Week 72
Population: Per Protocol (PP) population. Number of participants analyzed=participants with available data for specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 71
units on a scale | 7.3 (10.9)
Statistical Analysis 1: Comparison: Tocilizumab; Test type: Superiority or Other; p < 0.0001, Paired sample T-test

15. Primary Outcome: Change From Baseline in FACIT Fatigue Score at Week 96 in PP Population
Description: as for outcome 1
Time Frame: Baseline, Week 96
Population: Per Protocol (PP) population. Number of participants analyzed=participants with available data for specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 83
units on a scale | 7.3 (10.4)
Statistical Analysis 1: Comparison: Tocilizumab; Test type: Superiority or Other; p < 0.0001, Paired sample T-test

16. Secondary Outcome: Change From Baseline in SJC At Weeks 24, 48, 72, and 96
Description: 66 joints were assessed for swelling and joints are classified as swollen/not swollen giving a total possible swollen joint count score of 0 to 66. A negative change from baseline indicated improvement.
Time Frame: Baseline; Weeks 24, 48, 72 and 96
Population: ITT population. Here, 'n' signifies the number of participants with available data at specified timepoints.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 145
swollen joints
  Baseline (n=145) | 11.0 (6.6)
  Change From Baseline at Week 24 (n=124) | -7.3 (6.7)
  Change From Baseline at Week 48 (n=99) | -7.3 (6.4)
  Change From Baseline at Week 72 (n=79) | -7.6 (6.8)
  Change From Baseline at Week 96 (n=84) | -7.8 (6.8)
Statistical Analysis 1: Comparison: Tocilizumab; Change from baseline at Week 24; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: Tocilizumab; Change from baseline at Week 48; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test
Statistical Analysis 3: Comparison: Tocilizumab; Change from baseline at Week 72; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test
Statistical Analysis 4: Comparison: Tocilizumab; Change from baseline at Week 96; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test

17. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 20, ACR50 and ACR70 Response at Weeks 24, 48, 72, and 96
Description: ACR20 response: ≥20% improvement in TJC; ≥20% improvement in SJC; and ≥20% improvement in at least 3 of 5 remaining ACR core measures: Patient Assessment of Pain; Patient Global Assessment of Disease Activity (PtGA); Physician Global Assessment of Disease Activity (PGA); self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ-DI]); and either CRP or ESR. ACR50 response required ≥50% improvement in the above criteria and ACR70 response required ≥70% improvement in the above criteria.
Time Frame: Weeks 24, 48, 72 and 96
Population: as for outcome 3
Measure: Number; unit: percentage of partcipants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 121
percentage of partcipants
  ACR20: Week 24 (n=121) | 48.8
  ACR20: Week 48 (n=96) | 63.5
  ACR20: Week 72 (n=76) | 60.5
  ACR20: Week 96 (n=81) | 58.0
  ACR50: Week 24 (n=121) | 24.8
  ACR50: Week 48 (n=96) | 28.1
  ACR50: Week 72 (n=76) | 34.2
  ACR50: Week 96 (n=81) | 35.8
  ACR70: Week 24 (n=121) | 11.6
  ACR70: Week 48 (n=96) | 15.6
  ACR70: Week 72 (n=76) | 21.1
  ACR70: Week 96 (n=81) | 21.0

18. Secondary Outcome: Change From Baseline in Hemoglobin at Weeks 20, 44, 72 and 96
Time Frame: Baseline; Weeks 20, 44, 72 and 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: gram per deciliter
Arm/Group | Tocilizumab
Number analyzed (Participants) | 138
gram per deciliter
  Baseline (n=138) | 12.4 (1.4)
  Change From Baseline at Week 20 (n=122) | 0.7 (1.0)
  Change From Baseline at Week 44 (n=91) | 1.2 (1.2)
  Change From Baseline at Week 72 (n=73) | 1.0 (1.1)
  Change From Baseline at Week 96 (n=80) | 1.2 (1.3)

19. Secondary Outcome: C-reactive Protein Level
Time Frame: Baseline; Weeks 8, 16, 24, 36 48, 72 and 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligram per deciliter
Arm/Group | Tocilizumab
Number analyzed (Participants) | 133
milligram per deciliter
  Baseline (n=133) | 2.8 (5.6)
  Week 8 (n=114) | 0.3 (1.2)
  Week 16 (n=116) | 0.3 (0.6)
  Week 24 (n=112) | 0.2 (0.6)
  Week 36 (n=87) | 0.3 (0.8)
  Week 48 (n=89) | 0.2 (0.3)
  Week 72 (n=64) | 0.2 (0.6)
  Week 96 (n=75) | 0.5 (1.1)

20. Secondary Outcome: Erythrocyte Sedimentation Rate
Time Frame: Baseline; Weeks 8, 16, 24, 36 48, 72 and 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeter per hour
Arm/Group | Tocilizumab
Number analyzed (Participants) | 138
millimeter per hour
  Baseline (n=138) | 45.3 (27.1)
  Week 8 (n=125) | 10.6 (11.6)
  Week 16 (n=122) | 11.3 (14.9)
  Week 24 (n=118) | 8.8 (8.8)
  Week 36 (n=99) | 9.8 (12.0)
  Week 48 (n=96) | 8.3 (10.7)
  Week 72 (n=76) | 9.0 (9.5)
  Week 96 (n=74) | 7.4 (8.4)

21. Secondary Outcome: Participant Assessment of Pain (VAS)
Description: The mean score of pain as assessed by participants using a 100-mm horizontal VAS, where the left endpoint (0) indicated "No pain," and the right endpoint (100) indicated "Unbearable pain". Higher score indicated higher pain.
Time Frame: Baseline; Weeks 8, 16, 24, 36 48, 72 and 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 143
mm
  Baseline (n=143) | 70.3 (22.3)
  Week 8 (n=136) | 51.6 (26.7)
  Week 16 (n=132) | 53.0 (28.5)
  Week 24 (n=123) | 49.4 (26.8)
  Week 36 (n=104) | 44.7 (28.5)
  Week 48 (n=100) | 46.3 (28.8)
  Week 72 (n=76) | 42.3 (27.9)
  Week 96 (n=82) | 44.9 (28.0)

22. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) at Weeks 24, 48, 72, and 96
Description: HAQ: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline; Weeks 24, 48, 72 and 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 138
units on a scale
  Baseline (n=138) | 1.8 (0.7)
  Change From Baseline at Week 24 (n=112) | -0.4 (0.6)
  Change From Baseline at Week 48 (n=92) | -0.4 (0.6)
  Change From Baseline at Week 72 (n=73) | -0.4 (0.6)
  Change From Baseline at Week 96 (n=81) | -0.5 (0.6)

ADVERSE EVENTS:
Time Frame: From baseline up to 4 weeks after last dose of the study medication (up to Week 100)
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 36/145
Other Adverse Events (participants affected / at risk) | 134/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=145)
Angina unstable (Cardiac disorders) | 1
Myocardial infarction (Acute myocardial infarction and Myocardial infarction) (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Duodenitis (Gastrointestinal disorders) | 1
Gastric fistula (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 2
Pelvic mass (General disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 2
Otitis media chronic (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase/Aspartate aminotransferase elevations (Investigations) | 2
Catheterization cardiac (Investigations) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Erysipelas (Skin and subcutaneous tissue disorders) | 1
Cataract operation (Surgical and medical procedures) | 1
Cystocele repair (Surgical and medical procedures) | 1
Hernia repair (Surgical and medical procedures) | 1
Hysterectomy (Surgical and medical procedures) | 1
Lens extraction (Surgical and medical procedures) | 1
Obesity surgery (Surgical and medical procedures) | 1
Type IV hypersensitivity reaction (Immune system disorders) | 1
Hypertension (Vascular disorders) | 1
Rectal hemorrhage (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=145)
Leukopenia (Blood and lymphatic system disorders) | 32
Neutropenia (Blood and lymphatic system disorders) | 12
Upper respiratory tract infection (Infections and infestations) | 25
Viral Infection (Infections and infestations) | 14
Urinary tract infection (Infections and infestations) | 11
Nasopharyngitis (Infections and infestations) | 9
Alanine aminotransferase/Aspartate aminotransferase elevations (Investigations) | 47
Hyperlipidaemia (Metabolism and nutrition disorders) | 9
Exacerbation of rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 12
Headache (Nervous system disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 8
Nausea and Vomiting (Gastrointestinal disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.